CLINICAL TRIAL: NCT03744988
Title: Serum Androgen Levels as a Marker for the Severity of Preeclampsia
Status: Unknown | Type: Observational
Last Known Status: Active, not recruiting
Sponsor: Ain Shams University (Other)
Responsible Party: Principal Investigator, Joseph Adel Ibrahiem Johny, Principal Investigator, Ain Shams University
Other Study IDs: Joseph Adel Ibrahiem Johny
Record Dates: First submitted 2018-11-15; First posted 2018-11-19 (Actual); Last update posted 2018-11-20 (Actual); Status verified 2018-11

CONDITIONS: Severe Preeclampsia
MeSH Terms: conditions — Pre-Eclampsia

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 1 Week
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- control group: serum androgen levels will be measured in 25 normotensive pregnant women
  Interventions: Diagnostic Test: serum androgen levels
- mild preeclampsia: serum androgen levels will be measured in 25 mild preeclamptic patients
  Interventions: Diagnostic Test: serum androgen levels
- severe preeclampsia: serum androgen levels will be measured in 25 severe preeclamptic patients
  Interventions: Diagnostic Test: serum androgen levels

INTERVENTIONS:
Diagnostic Test: serum androgen levels — measurement of serum free and total testosterone

SUMMARY:
this study will be conducted to confirm the hypothesis of the previous studies and to list the high androgen levels as a precipitating factor for preeclampsia

DETAILED DESCRIPTION:
hypertensive disorders are one of the most important complications during pregnancy, which in combination with hemorrhage and infections make a dangerous triad, making them the major cause of maternal morbidity and mortality in 3.7-5% of all pregnancies.

Hypertensive disorders during pregnancy are classified into 4 categories, as recommended by the National High Blood Pressure Education Program Working Group on High Blood Pressure in Pregnancy:

* Chronic hypertension
* Preeclampsia-eclampsia
* Preeclampsia superimposed on chronic hypertension
* Gestational hypertension (transient hypertension of pregnancy or chronic hypertension identified in the latter half of pregnancy). This terminology is preferred over the older but widely used term "pregnancy-induced hypertension" (PIH) because it is more precise .

In 2008, the Society of Obstetricians and Gynecologists of Canada (SOGC) released revised guidelines that simplified the classification of hypertension in pregnancy into 2 categories, preexisting or gestational, with the option to add "with preeclampsia" to either category if additional maternal or fetal symptoms, signs, or test results support this .

Chronic hypertension is defined as blood pressure exceeding 140/90 mm Hg before pregnancy or before 20 weeks' gestation. When hypertension is first identified during a woman's pregnancy and she is at less than 20 weeks' gestation, blood pressure elevations usually represent chronic hypertension.

In contrast, new onset of elevated blood pressure readings after 20 weeks' gestation mandates the consideration and exclusion of preeclampsia .

Chronic Hypertension Chronic hypertension is a primary disorder in 90-95% of cases and may be either essential (90%) or secondary to some identifiable underlying disorder, such as renal parenchymal disease (eg, polycystic kidneys, glomerular or interstitial disease), renal vascular disease (eg, renal artery stenosis, fibro-muscular dysplasia), endocrine disorders (eg, adreno-corticosteroid or mineralocorticoid excess, pheochromocytoma, hyperthyroidism or hypothyroidism, growth hormone excess, hyperparathyroidism), coarctation of the aorta, or oral contraceptive use. About 20-25% of women with chronic hypertension develop preeclampsia during pregnancy .

Chronic hypertension occurs in up to 22% of women of childbearing age, with the prevalence varying according to age, race, and body mass index. Population-based data indicate that approximately 1% of pregnancies are complicated by chronic hypertension, 5-6% by gestational hypertension without proteinuria, and 1-2% by preeclampsia .

Differential Diagnosis

* Antiphospholipid Antibody Syndrome and Pregnancy
* Antithrombin Deficiency
* Aortic Coarctation
* Autoimmune Thyroid Disease and Pregnancy
* Cardiomyopathy, Peri-partum
* Common Pregnancy Complaints and Questions
* Cushing Syndrome
* Diabetes Mellitus and Pregnancy
* Disseminated Intravascular Coagulation
* Eclampsia
* Encephalopathy, Hypertensive
* Fetal Growth Restriction
* Gastrointestinal Disease and Pregnancy
* Glomerulonephritis, Acute
* Glomerulonephritis, Chronic
* Graves' Disease
* Hashimoto Thyroiditis
* Hematologic Disease and Pregnancy
* Hemolytic-Uremic Syndrome
* Hydatidiform Mole
* Hyper-aldosteronism, Primary
* Hyperparathyroidism
* Hypertension
* Hypertension, Malignant
* Hyperthyroidism
* Hypothyroidism
* Nephrotic Syndrome
* Normal Labor and Delivery
* Preeclampsia
* Protein C Deficiency
* Protein S Deficiency
* Pulmonary Disease and Pregnancy
* Systemic Lupus Erythematosus
* Systemic Lupus Erythematosus and Pregnancy
* Teratology and Drug Use During Pregnancy
* Thrombotic Thrombocytopenic Purpura Gestational Hypertension Gestational hypertension refers to hypertension with onset in the latter part of pregnancy (>20 weeks' gestation) without any other features of preeclampsia, and followed by normalization of the blood pressure postpartum. Of women who initially present with apparent gestational hypertension, about one third develops the syndrome of preeclampsia. As such, these patients should be observed carefully for this progression. The pathophysiology of gestational hypertension is unknown, but in the absence of features of preeclampsia, the maternal and fetal outcomes are usually normal .

Gestational hypertension may, however, be a harbinger of chronic hypertension later in life Furthermore, hypertension before pregnancy or during early pregnancy is associated with a twofold increased risk of gestational diabetes mellitus. Transient hypertension of pregnancy (ie, the development of isolated hypertension in a woman in late pregnancy without other manifestations of preeclampsia) is associated strongly with later development of chronic hypertension .

Although maternal diastolic blood pressure greater than 110 mm Hg is associated with an increased risk for placental abruption and fetal growth restriction, superimposed pre-eclamptic disorders cause most of the morbidity due to chronic hypertension during pregnancy .

Preeclampsia is defined as the new onset of hypertension and either proteinuria or end organ dysfunction after 20 weeks of gestation in a previously normotensive woman. In 2013, the American College of Obstetricians and Gynecologists removed proteinuria as an essential criterion for diagnosis of preeclampsia. They also removed massive proteinuria (5 grams/24hours) and fetal growth restriction as possible features of severe disease because massive proteinuria has a poor correlation with outcome and fetal growth restriction is managed similarly whether or not preeclampsia is diagnosed. Oliguria was also removed as a characteristic of severe disease.

Hypertension before 20 weeks' gestation is almost always due to chronic hypertension; new-onset or worsening hypertension after 20 weeks' gestation should lead to a careful evaluation for manifestations of preeclampsia .

Signs suggesting a secondary medical cause of chronic hypertension Centripetal obesity, "buffalo hump," and/or wide purple abdominal striae suggest glucocorticoid excess; other clinical signs may demonstrate hyperthyroidism, hypothyroidism, or growth hormone excess. In addition, a systolic bruit heard over the abdomen or in the flanks suggests renal artery stenosis, whereas radio femoral delay or diminished pulses in the lower versus upper extremities suggests coarctation of the aorta .

Women with chronic hypertension in pregnancy should be monitored for the development of worsening hypertension and/or the development of superimposed pre-eclampsia (the risk is approximately 25%). Laboratory investigations for pre-eclampsia should be repeated if the patient's blood pressure increases or if she develops signs or symptoms of preeclampsia .

ELIGIBILITY:
Inclusion Criteria:

* Pregnant women (primigravidas).
* Age between 20 and 35 years old.
* Live fetus.

Exclusion Criteria:

* Women younger than 20 years old and older than 35 years old
* Intrauterine fetal death.
* History of pre-gestational hypertension.
* History of hormonal disorders (thyroid gland disorders and hyperprolactinemia).
* Smoker.
* Polycystic ovary syndrome.
* Signs or symptoms of hyper-androgenism (hirsutism, acne, oily skin, etc.).
* Diabetes mellitus.
* Drug use except ordinary supplementation (iron, folic acid).

Ages: 20 Years to 35 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: patients will be divided into 3 groups
  1. control group : 25 normotensive pregnant women
  2. mild preeclampsia: 25 mild preeclamptic patients
  3. severe preeclampsia : 25 severe preeclamptic patients
Sampling Method: Non-Probability Sample
Enrollment: 75 (Actual)
Dates: Start 2017-10-01 (Actual); Primary Completion 2018-06-30 (Actual); Study Completion 2019-04-30 (Estimated)

PRIMARY OUTCOMES:
serum androgen levels as a marker for the severity of preeclampsia | 1 week
  assess if serum androgen levels could be used as a marker for the severity of preclampsia

CONTACTS AND LOCATIONS:
Overall Officials: Joseph A Ibrahiem, student, Principal Investigator — Ain Shams University
Locations (2):
- Egypt (2):
  - Ain Shams University, Cairo
  - AinShams University, Cairo

IPD SHARING:
Plan to Share IPD: Undecided
serum androgen levels as marker for the severity of preeclampsia